CLINICAL TRIAL: NCT04016727
Title: Variation in Rate of Orthodontic Tooth Movement in Response to Platelet Rich Plasma Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Armed Forces Institute of Dentistry, Pakistan (Other)
Responsible Party: Principal Investigator, Fatima Hamid, principal investigator, Armed Forces Institute of Dentistry, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: platelet rich plasma
Record Dates: First submitted 2019-06-28; First posted 2019-07-11 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Tooth Movement
Keywords: tooth movement; platelet rich plasma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP group (Experimental): patients in which 60 units of prp was injected
  Interventions: Biological: platelet rich plasma
- Control group (No Intervention): patients not given any intervention

INTERVENTIONS:
Biological: platelet rich plasma — Platelet rich plasma was prepared using patients own blood. 60 units of PRP was injected on one side of the arch using insulin syringe. Each patient served as his/her own control (the side with PRP injected) and experimental group (the side without PRP injected). Whether the right or left side served as control or experimental was determined by lottery method. Patients were recalled after 4 weeks and the measurements were repeated again between lateral incisors and canines at mid, cervical and incisal of the teeth and their mean was recorded.
  Arms: PRP group

SUMMARY:
PRP from 5 ml blood was prepared and 60 units were injected into the buccal vestibule of patient before initiating canine retraction using NiTi coil spring. Pre and post cervical, incisal and mid distances were measured using Vernier calliper.

DETAILED DESCRIPTION:
Platelet rich plasma was prepared using patients own blood. The production of PRP began with a 6-mL homologous blood sample that was withdrawn from the donor via venupuncture. One milliliter of the blood sample was set apart to determine the concentration of platelets and leukocytes in whole blood. The remaining 5 mL was mixed with an anticoagulant (3.8%, 1-mL sodium citrate) to prevent clotting. The blood sample was centrifuged at 113 g for 5 minutes to separate the plasma containing the platelets from the red cells. The plasma was drawn off the top and centrifuged for an additional 2 minutes at 3772 g to separate the platelets. Suitable platelet concentrations were achieved by the resuspension of PRP with plasma (high platelet concentration, 5 times the concentration in whole blood).

ELIGIBILITY:
Inclusion Criteria:

* patients requiring first premolar extractions

Exclusion Criteria:

* patients taking any drugs, steroids, NSAIDs and antibiotics
* patients with any co morbid conditions

Ages: 11 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2019-03-02 (Actual); Study Completion 2020-02-02 (Estimated)

PRIMARY OUTCOMES:
canine movement in mili meters | 1 month
  distance was measured using vernier caliper at mid cervical and incisal region

CONTACTS AND LOCATIONS:
Overall Officials: sana tariq, BDS, Study Chair — AFID rawalpindi
Locations (1):
- AFID, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No